CLINICAL TRIAL: NCT06529315
Title: Effects of Point-of-Care Ultrasound in Multidisciplinary Medical Wards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical Associate Professor, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 202405109RINA
Record Dates: First submitted 2024-07-08; First posted 2024-07-31 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Point-of-care Ultrasound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PoCUS (Experimental): Participants assigned to Group PoCUS will undergo point-of-care ultrasound evaluations by nurse practitioners/physicians within their first 24 hours of admission to the general ward.
  Interventions: Other: Point-of-Care Ultrasound
- Group Usual Care (No Intervention): Participants assigned to Group Usual Care will receive usual standard care.

INTERVENTIONS:
Other: Point-of-Care Ultrasound — The investigators will use point-of-care ultrasound to exam participants including lungs, heart, liver, spleen, kidney and bladder, etc.
  Arms: Group PoCUS

SUMMARY:
Point-of-care ultrasound (POCUS) is a bedside portable ultrasound technique utilized by healthcare providers to offer rapid and non-invasive diagnostic imaging. POCUS has proven particularly effective in critical care and emergency settings. However, its application in general medical wards, where patients often present with multiple comorbidities, remains under-researched. Additionally, the feasibility of nurse practitioners (NPs) performing POCUS is promising. Despite limited research on POCUS by less experienced operators, NP-conducted POCUS could provide timely, high-quality care, especially in situations with limited physician availability. The routine use of POCUS in patient admissions to medical wards may improve diagnostic accuracy, reduce diagnostic resource utilization, and shorten hospital stays.

DETAILED DESCRIPTION:
Point-of-care ultrasound (POCUS) is a bedside portable ultrasound technique utilized by healthcare providers to offer rapid and non-invasive diagnostic imaging. This method significantly aids in diagnosis and treatment by enhancing accuracy, guiding treatment adjustments, aiding procedural interventions, and reducing the time to appropriate treatment, ultimately leading to better patient outcomes. POCUS also decreases the reliance on other imaging modalities, providing real-time information and minimizing additional imaging needs.

POCUS has proven particularly effective in critical care and emergency settings. However, its application in general medical wards, where patients often present with multiple comorbidities, remains under-researched. The potential value of POCUS in these wards is notable, as it can facilitate early complication detection and timely treatment adjustments, reducing complication incidences.

Additionally, the feasibility of nurse practitioners (NPs) performing POCUS is promising. NPs, as frontline healthcare professionals, can use POCUS to enhance diagnostic and therapeutic capabilities. Despite limited research on POCUS by less experienced operators, NP-conducted POCUS could provide timely, high-quality care, especially in situations with limited physician availability. The routine use of POCUS in patient admissions to medical wards may improve diagnostic accuracy, reduce diagnostic resource utilization, and shorten hospital stays.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 years or older
2. Admitted directly from emergency department

Exclusion criteria:

1. End-of-life care
2. Immediate need for life-support therapy or ICU transfer
3. Airborne isolation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Proportion of accurate diagnosis | At 48 hours after admission to medical wards
  The proportion of accurate physician diagnosis achieved at 48 hours after admission to medical wards

SECONDARY OUTCOMES:
Hospital mortality | Until death, hospital discharge or up to 28 days
  Rate of hospital mortality of the participants
Rate of ICU transfer | Within 7 days after admission to medical wards
  Rate of participants requiring ICU care
Length of hospital stay | Until death, hospital discharge or up to 28 days
  The length of hospital stay of the participants
Categories and numbers of invasive procedures | Within 7 days after admission to medical wards
  Categories and numbers of invasive procedures required by the participants
Categories and numbers of imaging studies | Within 7 days after admission to medical wards
  The requests for additional categories and numbers of imaging studies for the participants

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ta Huang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zieleskiewicz L, Lopez A, Hraiech S, Baumstarck K, Pastene B, Di Bisceglie M, Coiffard B, Duclos G, Boussuges A, Bobbia X, Einav S, Papazian L, Leone M. Bedside POCUS during ward emergencies is associated with improved diagnosis and outcome: an observational, prospective, controlled study. Crit Care. 2021 Jan 22;25(1):34. doi: 10.1186/s13054-021-03466-z. PMID 33482873
- [Background] Ben-Baruch Golan Y, Sadeh R, Mizrakli Y, Shafat T, Sagy I, Slutsky T, Kobal SL, Novack V, Fuchs L. Early Point-of-Care Ultrasound Assessment for Medical Patients Reduces Time to Appropriate Treatment: A Pilot Randomized Controlled Trial. Ultrasound Med Biol. 2020 Aug;46(8):1908-1915. doi: 10.1016/j.ultrasmedbio.2020.03.023. Epub 2020 May 16. PMID 32430108
- [Background] Arvig MD, Lassen AT, Gaede PH, Gartner SW, Falster C, Skov IR, Petersen HO, Posth S, Laursen CB. Impact of serial cardiopulmonary point-of-care ultrasound exams in patients with acute dyspnoea: a randomised, controlled trial. Emerg Med J. 2023 Oct;40(10):700-707. doi: 10.1136/emermed-2022-212694. Epub 2023 Aug 18. PMID 37595984
- [Background] Patel S, Green A, Ashokumar S, Hoke A, Rachoin JS. Objective Methods of Assessing Fluid Status to Optimize Volume Management in Kidney Disease and Hypertension: The Importance of Ultrasound. J Clin Med. 2023 Oct 5;12(19):6368. doi: 10.3390/jcm12196368. PMID 37835014
- [Background] Pontet J, Yic C, Diaz-Gomez JL, Rodriguez P, Sviridenko I, Mendez D, Noveri S, Soca A, Cancela M. Impact of an ultrasound-driven diagnostic protocol at early intensive-care stay: a randomized-controlled trial. Ultrasound J. 2019 Sep 30;11(1):24. doi: 10.1186/s13089-019-0139-2. PMID 31595353
- [Background] Zieleskiewicz L, Muller L, Lakhal K, Meresse Z, Arbelot C, Bertrand PM, Bouhemad B, Cholley B, Demory D, Duperret S, Duranteau J, Guervilly C, Hammad E, Ichai C, Jaber S, Langeron O, Lefrant JY, Mahjoub Y, Maury E, Meaudre E, Michel F, Muller M, Nafati C, Perbet S, Quintard H, Riu B, Vigne C, Chaumoitre K, Antonini F, Allaouchiche B, Martin C, Constantin JM, De Backer D, Leone M; CAR'Echo and AzuRea Collaborative Networks. Point-of-care ultrasound in intensive care units: assessment of 1073 procedures in a multicentric, prospective, observational study. Intensive Care Med. 2015 Sep;41(9):1638-47. doi: 10.1007/s00134-015-3952-5. Epub 2015 Jul 10. PMID 26160727
- [Background] Wang PH, Chen JY, Ling DA, Lee AF, Ko YC, Lien WC, Huang CH. Earlier point-of-care ultrasound, shorter length of stay in patients with acute flank pain. Scand J Trauma Resusc Emerg Med. 2022 Apr 21;30(1):29. doi: 10.1186/s13049-022-01017-1. PMID 35449010
- [Background] Riishede M, Lassen AT, Baatrup G, Pietersen PI, Jacobsen N, Jeschke KN, Laursen CB. Point-of-care ultrasound of the heart and lungs in patients with respiratory failure: a pragmatic randomized controlled multicenter trial. Scand J Trauma Resusc Emerg Med. 2021 Apr 26;29(1):60. doi: 10.1186/s13049-021-00872-8. PMID 33902667
- [Background] Mozzini C, Di Dio Perna M, Pesce G, Garbin U, Fratta Pasini AM, Ticinesi A, Nouvenne A, Meschi T, Casadei A, Soresi M, Cominacini L. Lung ultrasound in internal medicine efficiently drives the management of patients with heart failure and speeds up the discharge time. Intern Emerg Med. 2018 Jan;13(1):27-33. doi: 10.1007/s11739-017-1738-1. Epub 2017 Aug 12. PMID 28803375
- [Background] Fraleigh CDM, Duff E. Point-of-care ultrasound: An emerging clinical tool to enhance physical assessment. Nurse Pract. 2022 Aug 1;47(8):14-20. doi: 10.1097/01.NPR.0000841944.00536.b2. PMID 35877142
- [Background] Manno E, Navarra M, Faccio L, Motevallian M, Bertolaccini L, Mfochive A, Pesce M, Evangelista A. Deep impact of ultrasound in the intensive care unit: the "ICU-sound" protocol. Anesthesiology. 2012 Oct;117(4):801-9. doi: 10.1097/ALN.0b013e318264c621. PMID 22990179
- [Background] Bernier-Jean A, Albert M, Shiloh AL, Eisen LA, Williamson D, Beaulieu Y. The Diagnostic and Therapeutic Impact of Point-of-Care Ultrasonography in the Intensive Care Unit. J Intensive Care Med. 2017 Mar;32(3):197-203. doi: 10.1177/0885066615606682. Epub 2016 Jul 9. PMID 26423745
- [Background] Atkinson PR, Milne J, Diegelmann L, Lamprecht H, Stander M, Lussier D, Pham C, Henneberry R, Fraser JM, Howlett MK, Mekwan J, Ramrattan B, Middleton J, van Hoving DJ, Peach M, Taylor L, Dahn T, Hurley S, MacSween K, Richardson LR, Stoica G, Hunter S, Olszynski PA, Lewis DA. Does Point-of-Care Ultrasonography Improve Clinical Outcomes in Emergency Department Patients With Undifferentiated Hypotension? An International Randomized Controlled Trial From the SHoC-ED Investigators. Ann Emerg Med. 2018 Oct;72(4):478-489. doi: 10.1016/j.annemergmed.2018.04.002. Epub 2018 Jun 2. PMID 29866583
- [Background] Yamada T, Ehara J, Funakoshi H, Endo K, Kitano Y. Effectiveness of point of care ultrasound (POCUS) simulation course and skills retention for Japanese nurse practitioners. BMC Nurs. 2023 Jan 23;22(1):21. doi: 10.1186/s12912-023-01183-2. PMID 36691022
- [Background] Huang C, Morone C, Parente J, Taylor S, Springer C, Doyle P, Temin E, Shokoohi H, Liteplo A. Advanced practice providers proficiency-based model of ultrasound training and practice in the ED. J Am Coll Emerg Physicians Open. 2022 Jan 11;3(1):e12645. doi: 10.1002/emp2.12645. eCollection 2022 Feb. PMID 35036994
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Lee SH, Yun SJ. Diagnostic performance of emergency physician-performed point-of-care ultrasonography for acute appendicitis: A meta-analysis. Am J Emerg Med. 2019 Apr;37(4):696-705. doi: 10.1016/j.ajem.2018.07.025. Epub 2018 Jul 14. PMID 30017693